CLINICAL TRIAL: NCT03251703
Title: Effects of Ultrasound-Guided Suprascapular Pulsed Radiofrequency Therapy on Chronic Shoulder Pain
Brief Title: Ultrasound-Guided Suprascapular Pulsed Radiofrequency
Acronym: PRF
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Serbülent Gökhan BEYAZ, associate professor, Sakarya University
Other Study IDs: Sakaray University
Record Dates: First submitted 2017-08-13; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: PAIN, INTRACTABLE, Shoulder
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound-Guided Suprascapular Pulsed Radiofrequency . — The ultrasound-Guided Suprascapular Pulsed Radiofrequency was administered under operating room conditions while the patient was monitored in a sitting position.An ultrasound-guided 22 G 5-mm active-tip 100-mm radiofrequency needle (SC-K; Top Neuropole, Tokyo, Japan) was pushed forward towards the suprascapular notch until it passed the transverse scapular ligament using an in-plane approach.

SUMMARY:
Shoulder pain is the second most common musculoskeletal disease in adults, and it often becomes chronic due to treatment difficulties.

Pulsed radiofrequency (PRF) therapy has become increasingly popular in the treatment of chronic shoulder pain due to its long duration of action and non-destructive method.

DETAILED DESCRIPTION:
These patients lacked pain control despite systemic analgesics and conservative therapy and applied to our pain polyclinics for shoulder pain lasting at least 3 months.

The ultrasound-guided SSPRF was performed in those patients with a reduction of 50% or more VAS score and those that reported healing in the AROM in the diagnostic SNB.

The resting, motion and sleeping shoulder pain assessments of the patients were done using a visual analog scale (VAS). The shoulder joint function was assessed using the Shoulder Pain and Disability Index (SPADI) questionnaire and the active range of motion (AROM) of the joint was measured using a goniometer In this study, investigators aimed to reveal the effects of ultrasound-guided suprascapular PRF (SSPRF) therapy applied to patients with chronic shoulder pain on both shoulder pain and function.

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years of age or older who were diagnosed with at least one of the following: adhesive capsulitis of the shoulder (M75.0), rotator cuff syndrome (M75.1), and impingement syndrome of shoulder (M75.4) according to the ICD-10 classifications. These patients lacked pain control despite systemic analgesics and conservative therapy (like physiotherapy) and applied to our pain polyclinics for shoulder pain lasting at least 3 months.

Exclusion Criteria:

Patients with other diseases causing chronic pain, those with neuropathic pain, those who had undergone surgery on the same shoulder, those with an allergy history from local anesthesia, those with abnormal coagulation tests, and those with cardiac pacemakers were excluded from this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: shoulder pain lasting at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of The Efficacy of Ultrasound-Guided Suprascapular Pulsed Radiofrequency | 1 years
  Retroscopic study

IPD SHARING:
Plan to Share IPD: No